CLINICAL TRIAL: NCT06682182
Title: Tislelizumab Combined with SOX and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Gastric Cancer with Peritoneal Metastasis: a Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yan Shi, Chief Physician, Southwest Hospital, China
Other Study IDs: SYIO-02
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer with Peritoneal Metastasis
Keywords: Tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tislelizumab+SOX — OX: S-1 dosing based on body surface area (BSA): <1.25m², 40 mg bid orally, 1.25-<1.5m², 50 mg bid orally, ≥1.5m², 60mg bid orally, days 1-14; Q3W; Oxaliplatin 130mg/m² IV day 1, for a total of 6 cycles.
  Tislelizumab: 200mg IV, day 1, Q3W, for a total of 6 cycles. HIPEC: Docetaxel 75mg/m² in 3500ml normal saline, at 43°C for 60 minutes.

SUMMARY:
The clinical trial aims to assess the efficacy and safety of Tislelizumab combined with the SOX regimen and HIPEC in treating gastric cancer with peritoneal metastasis. The primary and secondary objectives are as follows:

Primary objective: To evaluate the surgical conversion rate in patients with gastric cancer peritoneal metastasis treated with systemic chemotherapy plus immune checkpoint inhibitors combined with HIPEC.

Secondary objectives: To assess the safety, overall survival (OS), progression-free survival, tumor regression rate, incidence of adverse reactions during treatment, postoperative adverse reaction rates, and treatment efficacy of the combination therapy.

Participants will:

Be willing to receive SOX plus Tislelizumab combined with HIPEC treatment (exposure group), undergo one session of HIPEC followed by SOX plus immune checkpoint inhibitors (two cycles) to achieve stable disease (SD), partial response (PR), or complete response (CR). Patients who can undergo surgery after the second exploration will receive surgery and HIPEC treatment. If surgery is not possible, the next treatment plan will be discussed in a multidisciplinary team (MDT) meeting. Patients with progressive disease (PD) will also have their next treatment plan discussed in an MDT meeting.

Be willing to receive SOX combined with HIPEC treatment (observation group), undergo one session of HIPEC followed by SOX (two cycles) to achieve SD, PR, or CR. Patients who can undergo surgery after the second exploration will receive surgery and HIPEC treatment. If surgery is not possible, the next treatment plan will be discussed in an MDT meeting. Patients with PD will also have their next treatment plan discussed in an MDT meeting.

Treatment details:

SOX: S-1 dosing based on body surface area (BSA): <1.25m², 40 mg bid orally, 1.25-<1.5m², 50 mg bid orally, ≥1.5m², 60mg bid orally, days 1-14; Q3W; Oxaliplatin 130mg/m² IV day 1, for a total of 6 cycles.

Tislelizumab: 200mg IV, day 1, Q3W, for a total of 6 cycles. HIPEC: Docetaxel 75mg/m² in 3500ml normal saline, at 43°C for 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed Her-2 negative gastric adenocarcinoma who have not received chemotherapy, radiotherapy, or other anti-cancer treatments before the start of the clinical trial.

Age between 18 to 80 years old, Eastern Cooperative Oncology Group (ECOG) performance status: 0-1.

American Joint Committee on Cancer (AJCC) 8th edition TNM staging of T1-4aNxM1 (limited to peritoneal metastasis or the presence of ascites beyond the pelvis), without obstruction, perforation, or bleeding risk.

Peritoneal Cancer Index (PCI) ≤ 20. Good bone marrow reserve function, with blood routine meeting the following conditions: white blood cell count ≥ 3×10^9/L, neutrophil count ≥ 1.5×10^9/L, platelet count ≥ 100×10^9/L, hemoglobin ≥ 90 g/L.

Good organ function, with biochemical tests meeting the following conditions: Alanine aminotransferase (ALT) ≤ 2.5× upper limit of normal (ULN), Aspartate aminotransferase (AST) ≤ 2.5× ULN, serum total bilirubin ≤ 1.5× ULN, blood creatinine ≤ 1.5× ULN or creatinine clearance ≥ 50 mL/min.

International Normalized Ratio (INR) ≤ 1.5, Prothrombin Time (PT) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN.

Urine protein < 2+, if urine protein ≥ 2+ then 24-hour urine protein quantification must show protein ≤ 1g.

Agreement to provide blood/tissue samples. Expected survival of more than 3 months. Female subjects agree to strict contraception; male subjects with partners of childbearing potential agree to use effective contraception during the study period.

Voluntary signing of the informed consent form, willingness and ability to comply with planned visits, study treatments, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Patients who are receiving other drug clinical trials or have participated in any drug clinical trials within one month before enrollment.

Other anti-tumor treatments (chemotherapy, radiotherapy, surgery, immunotherapy, biotherapy, chemoembolization) except for study medication. Palliative external irradiation for non-target lesions is allowed.

Prior use of similar chemotherapy drugs or immune checkpoint inhibitors. Presence of non-pelvic abdominal metastatic lesions in the liver, lungs, para-aortic lymph nodes, bones, brain, adrenal glands, etc.; patients with peritoneal metastasis in the small bowel mesentery (regions 9-12) must be excluded.

Gastrointestinal perforation, obstruction, or uncontrollable diarrhea within 6 months before enrollment.

Other untreated or concurrent tumors, except for cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumors. Patients may be enrolled if the tumor was cured and there has been no evidence of disease for more than 5 years. All other tumors must have been treated at least 5 years before enrollment.

Symptomatic meningioma. History of active autoimmune disease or refractory autoimmune disease. Received corticosteroids (>10mg/day prednisone or equivalent dose of steroids) or other systemic immunosuppressive therapy within 14 days before enrollment, excluding the following treatments: steroid hormone replacement therapy (≤10mg/day); local steroid therapy; and short-term prophylactic steroid therapy for allergy or nausea and vomiting.

History of HIV infection or active hepatitis B/C virus infection. Persistent > Grade 2 bacterial, fungal, viral, or other infections.

Active or clinically significant cardiac disease:

Congestive heart failure > New York Heart Association (NYHA) Class 2; Active coronary artery disease; Arrhythmias requiring treatment other than beta-blockers or digoxin; Unstable angina (angina symptoms at rest), new-onset angina within 3 months before enrollment, or new myocardial infarction with unhealed wounds, ulcers, or fractures within 6 months before enrollment.

Patients with renal failure requiring hemodialysis or peritoneal dialysis. Patients requiring medication for epilepsy. History of organ transplantation (including corneal transplants). Allergy or suspected allergy to the study medication or similar drugs. Pregnant or breastfeeding women. Major surgery, open biopsy, or major traumatic surgery within 4 weeks before recruitment (excluding biliary stents or percutaneous biliary drainage).

History of vaccination within 4 weeks before enrollment. Patients deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically confirmed Her-2 negative gastric adenocarcinoma who have not received chemotherapy, radiotherapy, or other anti-cancer treatments before the start of the clinical trial.American Joint Committee on Cancer (AJCC) 8th edition TNM staging of T1-4aNxM1 (limited to peritoneal metastasis or the presence of ascites beyond the pelvis), without obstruction, perforation, or bleeding risk.
  Peritoneal Cancer Index (PCI) ≤ 20.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Conversion surgery rate | 1 year
  Conversion surgery rate (the proportion of enrolled patients achieving R0 resection after treatment) for gastric cancer patients with peritoneal metastasis treated with Tislelizumab combined with HIPEC

IPD SHARING:
Plan to Share IPD: No